| Title | Natural History of Photoreceptor Degeneration Related to USH1b, Clinical Parameters, and Validation of Functional Vision Tests |
|---|---|
| Acronyme | МҮО7А |
| Principal Investigator | Pr. Isabelle AUDO |
| Sponsor | Hôpital National de la Vision des Quinze-Vingts, Paris (France) |
| | nherited retinal diseases (IRD) are a heterogeneous group of disorders that progressively lead to severe visual impairments with limited therapeutic options. Rod dystrophy, also known as retinitis pigmentosa (RP), is the most common form of IRD, with an estimated global prevalence of 1 in 4,500. Approximately 20 to 30% of rod-cone dystrophy cases are syndromic forms, among which Usher syndrome (USH) is the most frequent (estimated prevalence of 1 to 4 in 25,000), accounting for 50% of cases of combined deafness and blindness in males and 3 to 6% of all childhood deafness cases. |
| Justification for the Study | Type 1 Usher syndrome (USH1) is the most severe form of USH and typically presents with severe to profound congenital sensorineural deafness, vestibular areflexia, and early-onset rod-cone dystrophy (i.e., during the first decade of life). Mutations in nine genes have been associated with USH1, among which biallelic mutations in MYO7A represent 70% of cases. These specific mutations are known as USH1B syndrome. |
| | Currently, there is no treatment available for USH1B, representing a significant unmet medical need for this severe form of USH. |
| Study Objectives | <ol> <li>Study of the natural history of retinal degeneration in a large USH1B cohort</li> <li>Validation of functional vision tests based on virtual reality and two patient-reported questionnaires</li> </ol> |
| | Research with minimal risks and constraints, Category 2 |
| Study Category and Type | This is a prospective and longitudinal study focusing on the natural history and progression of inherited retinal diseases related to USH1b, as well as the validation of clinical parameters and functional vision tests. |
| | Functional Tests: |
| Evaluation Criteria and Parameters | <ul> <li>Letter score from Best-Corrected Visual Acuity (BCVA) using the Early Treatment Diabetic Retinopathy Study (ETDRS) scale</li> <li>In case of very low visual acuity: Berkeley Rudimentary Vision Test (BRVT)</li> <li>Low Luminance Visual Acuity (LLVA) using ETDRS or HOTV charts</li> <li>Color Contrast Sensitivity using the Lanthony 15-HUE test and Cambridge Colour Test</li> <li>Contrast Sensitivity with the backlit Pelli-Robson chart</li> </ul> |
| | <ul> <li>Mesopic Microperimetry (MAIA)</li> <li>Kinetic Visual Field testing (Octopus 900)</li> <li>Static Visual Field testing (Octopus 900)</li> </ul> |

Retinal Function evaluated by Full-Field Stimulus Threshold (FST) testing (global photoreceptor sensitivity) Retinal Function assessed by full-field electroretinogram (ERG) responses to rod- and cone-specific stimuli (measuring amplitude and peak time) **Structural Tests: Retinography** (Clarus) Fundus Autofluorescence (FAF) imaging using both short-wavelength autofluorescence (SWAF) and near-infrared autofluorescence (NIRAF) (HRA2) **Spectral Domain Optical Coherence Tomography (SD-OCT) Optical Coherence Tomography Angiography (OCT-A) Axial Length Measurements Objective Refraction and Non-contact Tonometry** Quality of Life: Responses to the two patient-reported outcome questionnaires: o The Michigan Vision-Related Anxiety Questionnaire (MAVQ): A <u>Psychosocial Outcomes Measure for Inherited Retinal</u> **Degenerations** o The Michigan Retinal Degeneration Questionnaire (MRDQ): A Patient-Reported Outcome Instrument for Inherited Retinal **Degenerations** Age ≥ 3 years Clinical diagnosis of Usher Syndrome Type 1 (USH1) in both eyes, defined as profound congenital deafness, vestibular dysfunction, and rod-cone dystrophy, with biallelic class 4 or 5 variants in the MYO7A gene Affiliation with, or beneficiary of, a social security system (according to article L1121-8-1 of the French Public Health Code) Additional Inclusion Criteria for Participants in the MOST-VR and VR-ViSA **Inclusion Criteria** (Streetlab) Tests: Sufficient understanding of spoken and signed French to ensure proper comprehension of the tasks and instructions Presence of a cochlear implant allowing for comprehension of auditory instructions during the virtual reality mobility test, with a Mini-Mental State Examination (MMSE) score  $\geq 20/25$ Age between 18 and 75 years Inability to attend or complete all study visits Anticipated participation in an experimental treatment trial at any point during the study Presence of ocular conditions that could impact retinal status other than **Exclusion Criteria** retinitis pigmentosa (e.g., history of retinal detachment, glaucoma, vein occlusion, diabetic retinopathy, etc.) Prior participation in the USH1B gene therapy trial (USHSTAT, NCT01505062) Pregnant, postpartum, or breastfeeding women (according to article L1121-5 of the French Public Health Code)

| | transfer and the second of the |
|---|---|
| | <ul> <li>Individuals deprived of liberty by judicial or administrative decision (according to article L1121-6 of the French Public Health Code)</li> <li>Adults under legal protection or unable to provide informed consent (according to article L1121-8 of the French Public Health Code)</li> </ul> |
| | - Additional Exclusion Criteria for Participants in the MOST-VR and VR-ViSA |
| | Tests: |
| | <ul> <li>MMSE score (visual items excluded) ≤ 20/25</li> <li>Physical or cognitive impairment likely to interfere with mobility</li> </ul> |
| | - Ongoing treatment with medications that may affect motor, visual, or |
| | cognitive function (e.g., antipsychotics, neuroleptics) or that may interfere with study assessments |
| | - Occurrence of other medical conditions or treatments likely to interfere with the assessments planned during the study. |
| Criteria for Early<br>Discontinuation or Study | <ul> <li>Voluntary withdrawal: A participant may decide to discontinue participation at any time, without justification and without affecting their future medical care.</li> </ul> |
| Withdrawal | - Investigator decision: A participant may also be withdrawn from the study at the discretion of the investigator, for reasons such as safety concerns, protocol non-compliance, or any other reason deemed appropriate. |
| Constraints and Risks | The procedures involved in this study may expose participants to the following medical risks: |
| | - Pupil dilation, performed as part of the ophthalmologic evaluation, may cause side effects, with a risk of acute angle-closure glaucoma estimated at less than 1 in 5000 cases. Risk factors will be systematically screened during the ophthalmologic examination, particularly through slit-lamp evaluation. |
| | <ul> <li>Placement of corneal electrodes for the full-field electroretinogram (ERG), as well as the instillation of topical anesthetic eye drops (oxybuprocaine), may occasionally cause corneal erosion or corneal edema, resulting in pain lasting 24 to 48 hours after the examination. This rare complication will be systematically assessed during the fundus examination, and a healing eye drop will be prescribed if necessary.</li> </ul> |
| | - Completion of patient-reported questionnaires may induce psychological side effects, such as increased anxiety or emotional stress. However, such reactions are typically transient, and participants are free to discontinue at any time if needed. |
| Population | A total of 60 participants are expected to be recruited for this study. The study is divided into three sub-cohorts: two pediatric cohorts (n=10 patients, ages 3–5 and 6–13 years) and one mixed adolescent and adult cohort (aged 14 and older n=50). |
| Research Procedure | See Tables 1, 2, and 3 The following procedures are not part of routine care and are therefore added specifically for the research: |
| | - MOST-VR and VR-ViSA tests (Streetlab) |

## **Protocol Summary**

| Projected Research<br>Timeline | <ul> <li>Planned Study Start Date: June 2025</li> <li>Duration of Participation per Participant: 4 years (48 months)</li> <li>Visit Frequency: 6 visits in total (initial visit, reproducibility visit, and 4 follow-up visits)</li> <li>Planned Enrollment Period: 6 months. If recruitment goals are not met within this timeframe, the enrollment period may be extended up to a total of 24 months.</li> <li>Total Study Duration: 72 months (48 months participation + up to 24 months enrollment extension)</li> </ul> |
|---|---|
| Funding Source | Foundation Fighting Blindness |
| Reimbursement of Expenses | The study will cover the costs of all examinations beyond standard care, including contrast sensitivity, color contrast vision, mesopic microperimetry, FST, and SS-OCT-A. Additionally, travel and accommodation expenses related to these visits will be reimbursed upon presentation of receipts and prior approval for each evaluation visit. |

Table 1. Test Protocol for the Pediatric Cohort Aged 3 to 5 Years

| Visits | Initial<br>visit<br>(D+0) | Reproductibility<br>visit (D+1 à D+30) | M12<br>± 3M | M24<br>± 3M | M36<br>± 3M | M48<br>± 3M | Duration<br>of the<br>examinati<br>on<br>(minutes) |
|---|---|---|---|---|---|---|---|
| Procedures and tests | | | | | | | |
| Informed Consent | Х | - | - | - | - | - | 15 |
| Demographics / Medical History | Х | - | Х | Х | Х | Х | 10 |
| Concomitant Medications /<br>Adverse Events | Х | - | Х | Х | Х | Х | 5 |
| Objective Refraction + Air<br>Tonometry | Х | - | Х | Х | х | Х | 5 |
| Axial Length Measurement | Х | - | Χ | Х | Χ | Χ | 5 |
| Visual Acuity Measurement | Х | - | Χ | Χ | Χ | Χ | 15 |
| Full-Field Electroretinogram (ERG) | Х | - | Х | Х | Х | Х | 60 |
| Ophthalmological Examination | Х | - | Х | Х | Х | Х | 5 |
| Retinal Photography | Х | | Х | Х | Х | Х | 10 |
| Blue and Near-Infrared Fundus<br>Autofluorescence Imaging<br>(HRA2, 30° and 50°) | Х | - | Х | Х | Х | Х | 15 |
| Spectral-Domain and Swept-<br>Source Optical Coherence<br>Tomography (SD-OCT and OCT-<br>Angiography) | Х | - | Х | Х | Х | х | 25 |

<sup>&</sup>lt;sup>1</sup> The full-field electroretinogram (ERG) will not be performed if previous data showed no detectable response.

<sup>&</sup>lt;sup>2</sup> Axial length measurement may be difficult to perform in some subjects depending on their level of concentration.

Table 2. Testing protocol for the pediatric cohort aged 6 to 13 years

| Visits | Initial<br>visit<br>(D+0) | Reproductibility<br>visit (D+1 à D+30) | M12<br>± 3M | M24<br>± 3M | M36<br>± 3M | M48<br>± 3M | Duration<br>of the<br>examinati<br>on<br>(minutes) |
|---|---|---|---|---|---|---|---|
| Procedures and tests | | | | | | | |
| Informed Consent | Х | - | - | - | - | - | 15 |
| Demographics / Medical History | Х | - | Х | Х | Х | Х | 10 |
| Concomitant Medications /<br>Adverse Events | Х | - | X | Х | Х | Х | 5 |
| Objective Refraction + Air<br>Tonometry | Х | - | Х | Х | Х | Х | 5 |
| Axial Length Measurement <sup>2</sup> | Χ | <u>-</u> | Χ | Χ | Χ | Χ | 5 |
| Best Corrected Visual Acuity (ETDRS or BRVT) | Х | - | Х | Х | Х | Х | 15 |
| Low Luminance Best Corrected<br>Visual Acuity (LLVA) | Х | - | Х | Х | Х | Х | 10 |
| Color Contrast Sensitivity (15<br>HUE Lanthony Test) | Х | - | Х | Х | Х | Х | 30 |
| Contrast Sensitivity (Pelli-<br>Robson) | Х | - | Х | Х | Х | Х | 15 |
| Kinetic Visual Field (Octopus 900) | Х | - | Х | Х | Х | Х | 45 |
| Full-field Electroretinogram (ERG) <sup>1</sup> | Х | - | Х | Х | Х | Х | 60 |
| Ophthalmological Examination | Х | - | Χ | Χ | Х | Х | 5 |
| Retinophotography | Χ | - | Χ | Χ | Χ | Χ | 10 |
| Blue and Near-Infrared Fundus<br>Autofluorescence (HRA2, 30°<br>and 50°) | X | - | X | X | X | Х | 15 |
| Spectral-Domain and Swept-<br>Source Optical Coherence<br>Tomography (SD-OCT and SS-<br>OCT-A) | Х | - | Х | X | Х | х | 25 |

<sup>&</sup>lt;sup>1</sup> L'électrorétinogramme plein champ ne sera pas effectué si les données antécédentes n'ont montré aucune réponse détectable.

<sup>&</sup>lt;sup>2</sup> La mesure de la longueur axiale peut être difficilement réalisée chez certains sujets en fonction de leur concentration

**Table3.** Test Protocol for the Adolescent (≥14 years) and Adult Cohort

| Visits | Initial visit<br>(D+0) | Reproductibility<br>visit (D+1 à D+30) | M12<br>± 3M | M24<br>± 3M | M36<br>± 3M | M48<br>± 3M | Duration of<br>the<br>examination<br>(minutes) |
|---|---|---|---|---|---|---|---|
| Procedures and tests | | | | | | | (minutes) |
| Informed Consent | X | - | - | - | - | - | 15 |
| Demographics / Medical History | X | - | X | X | X | X | 10 |
| Concomitant Medications / | 37 | | 37 | v | N/ | 37 | 5 |
| Adverse Events | X | - | X | X | X | X | 5 |
| Objective Refraction + Air | X | | X | X | X | X | 5 |
| Tonometry | Λ | <u>-</u> | Λ | Λ | Λ | Λ | 3 |
| Axial Length Measurement | X | - | X | X | X | X | 5 |
| Best Corrected Visual Acuity<br>(ETDRS or BRVT) | X | - | X | X | X | X | 15 |
| Low Luminance Best Corrected<br>Visual Acuity (LLVA) | X | - | X | X | X | X | 10 |
| Color Contrast Sensitivity<br>(Cambridge Color Test, Triverctor<br>protocol) | X | - | X | X | X | X | 30 |
| Contrast Sensitivity (Pelli-Robson) | X | - | X | X | X | X | 15 |
| Mesopic Microperimetry (MAIA) | X | X | X | X | X | X | 30 |
| Static Visual Field (Octopus 900) | X | - | X | X | X | X | 60 |
| Kinetic Visual Field (Octopus 900) | X | - | X | X | X | X | 45 |
| Full-field Stimulus Threshold (FST) | X | - | X | X | X | X | 90 |
| Full-field Electroretinogram (ERG) <sup>1</sup> | X | - | X | X | X | X | 60 |
| Ophthalmological Examination | X | - | X | X | X | X | 5 |
| Retinophotography | X | | X | X | X | X | 10 |
| Blue and Near-Infrared Fundus | | | | | | | |
| Autofluorescence (HRA2, 30° and 50°) | X | - | X | X | X | X | 15 |
| Spectral-Domain and Swept- | | | | | | | |
| Source Optical Coherence | X | - | X | X | X | X | 25 |
| Tomography (OCT and OCT-A) | | | | | | | |
| Patient-Reported Outcome | | | _ | _ | _ | _ | |
| Questionnaires (MVAQ and<br>MRDQ) | X | <u>-</u> | X | X | X | X | 30 |
| Streetlab Tests (MOST-VR, VR-<br>ViSA)² | X | X | | X | | | 150 |

<sup>1.</sup> The full-field electroretinogram (ERG) will not be performed if prior data showed no detectable response.

<sup>2.</sup> MOST-VR and VR-ViSA tests will only be conducted in participants aged 18 years and older who meet the inclusion criteria specified in the table "Inclusion Criteria for MOST-VR and VR-ViSA Tests."